CLINICAL TRIAL: NCT05743855
Title: The Effect of Co-therapy Chiropractic Plus Nutritional Supplement in Patients Experiencing Chronic Pain and Inflammation.
Brief Title: The Effect of Chiropractic Plus Nutritional Supplement in Patients With Chronic Pain and Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00032192
Record Dates: First submitted 2023-01-16; First posted 2023-02-24 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain; Inflammatory Response
MeSH Terms: conditions — Chronic Pain | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants consume 1 serving of Placebo daily and attend weekly chiropractor sessions for 12 weeks.
  Interventions: Other: Placebo
- Treatment Group (Experimental): Participants consume 1 serving of the Nutrional supplement daily and attend weekly chiropractor sessions for 12 weeks.
  Interventions: Dietary Supplement: Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement — Nutritional Supplement + Chiropract sessions
  Other Names: Chiropract sessions
  Arms: Treatment Group
Other: Placebo — Placebo + Chiropractic sessions
  Other Names: Chiropract sessions
  Arms: Placebo

SUMMARY:
Evaluating the effect of a combined therapy of chiropractic sessions plus nutritional supplement containing hemp, omega-3 fatty acids, and broccoli extract oil in patients experiencing chronic pain and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain (>3years)

Exclusion Criteria:

* GABA/opioid medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Pain level using the Brief Pain Inventory (BPI) after 12 weeks. | Baseline and 12 weeks
  The BPI is a validated self-reporting instrument assessing pain. Possible score range 0-10 with higher scores indicating higher pain levels. The instrument contains 9 items.
Change from baseline in Pain intensity using the 11-Point Numeric Rating Scale (11-NRS) after 12 weeks. | Baseline and 12 weeks
  The 11-NRS is a validated self-reporting instrument assessing pain level. Possible score ranges from '0' representing "no pain" to '10' representing "worst pain imaginable".

SECONDARY OUTCOMES:
Reactive oxygen species (ROS) status | At baseline and after 12 weeks
  Reactive oxygen species (ROS) status in the peripheral blood mononuclear cells was used to assess participant's inflammation biomarkers.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Randolph Chiropractic Health Center, Charlotte, North Carolina
  - Trull Chiropractic PA, Kannapolis, North Carolina
  - Combined Chiropractic & Acupuncture PLLC, Mooresville, North Carolina

IPD SHARING:
Plan to Share IPD: No